CLINICAL TRIAL: NCT03752411
Title: The Use of Nomi Technology to Monitor Opioid Use
Brief Title: Environment Analysis Inside an Investigational Prescription Bottle
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 18-0022
Record Dates: First submitted 2018-11-21; First posted 2018-11-26 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Chronic Pain
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Research Bottle (Experimental): This group will have medication dispensed in a research bottle.
  Interventions: Other: Research Bottle
- Regular prescription Bottle (Placebo Comparator): This group will have medication dispensed in a regular prescription bottle
  Interventions: Other: Regular prescription Bottle

INTERVENTIONS:
Other: Research Bottle — The purpose of the study is to test a research prescription bottle that will monitor the physical environment inside the bottle.
  Arms: Research Bottle
Other: Regular prescription Bottle — This will test if the research bottle changes behavior relative to the research bottle
  Arms: Regular prescription Bottle

SUMMARY:
The purpose of the study is to test a research prescription bottle that will monitor the physical environment inside the bottle.

DETAILED DESCRIPTION:
The purpose of the study is to test a research prescription bottle that will monitor the physical environment inside the bottle. The participant will be asked to keep the medication in the bottle and to remove each pill immediately before taking it.

The participant will not store medications in pill organizers, other pill bottles, pockets, purses, etc. The participant will keep a record of when the participant removes a pill from the bottle and takes it. Certain aspects of this study will be withheld from the participant to preserve the integrity of the study. This information will be revealed at the conclusion of the study.

ELIGIBILITY:
Inclusion Criteria:

* chronic pain > 3 months duration
* major source of pain is due to low back pain diagnosis
* prescribed only one type of opioid: hydrocodone 10mg/325 mg acetaminophen
* Last urine drug study was done between 6-12 months ago
* will have a return to clinic visit in 3 months

Exclusion Criteria:

* concurrent use of other opioids
* use of intrathecal device
* use of spinal cord stimulator
* presence of pain due to cancer, chemotherapy, radiation treatment and/or cancer related surgery
* dementia
* illiteracy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2022-11-05 (Actual); Study Completion 2023-11-05 (Actual)

PRIMARY OUTCOMES:
total medication dose | day 90
  pain medication dose (mg)
total Pain scale | day 90
  On a scale of 0-10 where 0 is no pain and 10 is the worst pain ever felt.
total nausea scale | day 90
  On a scale of 0-3 where 0=no nausea, 1= mild, 2= moderate, and 3= severe
total vomiting scale | day 90
  On a scale of 0-3 where 0=no vomiting, 1= mild, 2= moderate, and 3= severe
total sedation scale | day 90
  On a scale of 0-3 where 0=no sedation, 1= mild, 2= moderate, and 3= severe
total bowel movements | day 90
  number of bowel movements (whole number)
total type of bowel movement | day 90
  choose one of the following: hard, soft, loose
overall satisfaction with pain control | day 90
  0-10 scale where 0 is dissatisfied and 10 is very satisfied

SECONDARY OUTCOMES:
opioid related behavior in treatment questionnaire | day 90
  Measures opioid misuse score (number 0-40) where 0-10 is low misuse, 11-30 is moderate misuse and 31-40 is high misuse
prescribed opioids difficulty scale | day 90
  measures opioid management score (number 0-32) where 0-10 is low difficulty, 11-21 is moderate difficulty and 22-32 is high levels of difficulty
Barretts impulsivity questionnaire | day 90
  Measures impulsivity behavior core (number 0-120) where 0-40 is low levels of impulsivity, 41-80 is moderate levels of impulsivity, and 81-120 is high levels of impulsivity

CONTACTS AND LOCATIONS:
Overall Officials: Denise Wilkes, MD-PhD, Study Director — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Robinson-Papp J, George MC, Wongmek A, Nmashie A, Merlin JS, Ali Y, Epstein L, Green M, Serban S, Sheth P, Simpson DM. The Quantitative Analgesic Questionnaire: A Tool to Capture Patient-Reported Chronic Pain Medication Use. J Pain Symptom Manage. 2015 Sep;50(3):381-6. doi: 10.1016/j.jpainsymman.2015.03.013. Epub 2015 Apr 23. PMID 25912277
- [Derived] Houghton DC, Merritt CR, Miller SN, Mitchell JM, Parker D, Hommel JD, Cunningham KA, Wilkes DM. Electronic Real-Time Monitoring Reveals Limited Adherence to Long-Term Opioid Prescriptions in Pain Patients. J Pain Res. 2024 May 21;17:1815-1827. doi: 10.2147/JPR.S436898. eCollection 2024. PMID 38799276